CLINICAL TRIAL: NCT01084876
Title: A Double-blind, Randomised, Parallel Group, Phase III Study to Demonstrate Equivalent Efficacy and Comparable Safety of CT-P6 and Herceptin, Both in Combination With Paclitaxel, in Patients With Metastatic Breast Cancer
Brief Title: Demonstrate Efficacy and Safety of Metastatic Breast Cancer
Acronym: Compare
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-P6/3.1
Record Dates: First submitted 2010-03-09; First posted 2010-03-11 (Estimated); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Herceptin; metastatic breast cancer; CT-P6; Her 2-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — CT-P6; Trastuzumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-P6 & Paclitaxel (Experimental): CT-P6 was administered at a loading dose of 8 mg/kg body weight by intravenous (IV) infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 body surface area (BSA) as a continuous 3-hour IV infusion on the day following the first dose of study drug (CT-P6). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death or discontinuation.
  Interventions: Drug: CT-P6; Drug: Paclitaxel
- Herceptin & Paclitaxel (Active Comparator): Herceptin was administered at a loading dose of 8 mg/kg body weight by IV infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 BSA as a continuous 3-hour IV infusion on the day following the first dose of study drug (Herceptin). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death or discontinuation.
  Interventions: Drug: Herceptin; Drug: Paclitaxel

INTERVENTIONS:
Drug: CT-P6 — Administered every 3 weeks
  Arms: CT-P6 & Paclitaxel
Drug: Herceptin — Administered every 3 weeks
  Other Names: Trastuzumab
  Arms: Herceptin & Paclitaxel
Drug: Paclitaxel — Administered every 3 weeks

SUMMARY:
The purpose of the study is to demonstrate equivalence

DETAILED DESCRIPTION:
Patients will receive CT-P6 or Herceptin every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are females
* Have Her 2 over-expression
* Have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* Current clinical or radiographic evidence central nervous system (CNS) metastases
* Current Known infection
* Pregnant or nursing mother

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Investigational Site, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 475 patients initiated Main Study Treatment Period and were included in the Full Analysis Set (FAS).
Groups:
- CT-P6: CT-P6 was administered at a loading dose of 8 mg/kg body weight by intravenous (IV) infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 body surface area (BSA) as a continuous 3-hour IV infusion on the day following the first dose of study drug (CT-P6). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death or discontinuation.
- Herceptin: Herceptin was administered at a loading dose of 8 mg/kg body weight by IV infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 BSA as a continuous 3-hour IV infusion on the day following the first dose of study drug (Herceptin). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death or discontinuation.
Period: Main Study Treatment Period
Arm/Group | CT-P6 | Herceptin
Started (Patient disposition of the main study treatment period in the Phase 3 study (CT-P6 3.1) was analyzed in conjunction with that of the Phase 1/2b study (CT-P6 1.1).) | 244 | 231
Completed | 185 | 192
Not Completed | 59 | 39
Not completed — Adverse Event | 12 | 7
Not completed — Disease Progression | 41 | 24
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Other Reason | 0 | 1
Not completed — Other | 0 | 1
Period: Treatment Period Beyond Cycle 8
Arm/Group | CT-P6 | Herceptin
Started (Patient disposition of the treatment period beyond Cycle 8 in the Phase 3 study (CT-P6 3.1) was analyzed in conjunction with that of the Phase 1/2b study (CT-P6 1.1). Discontinuation reasons for patients who completed treatment at Cycle 8 and discontinued before starting Cycle 9 were also counted.) | 168 | 168
Completed | 0 | 0
Not Completed | 168 | 168
Not completed — Adverse Event | 8 | 2
Not completed — Disease Progression | 129 | 119
Not completed — Physician Decision | 6 | 5
Not completed — Withdrawal by Subject | 12 | 20
Not completed — Other Reason | 7 | 13
Not completed — Other | 6 | 9

BASELINE CHARACTERISTICS:
Population: All baseline characteristics of the Phase 3 study (CT-P6 3.1) listed below were analyzed in conjunction with those of the Phase 1/2b study (CT-P6 1.1).
Groups:
- CT-P6: CT-P6: 8 mg/kg for loading or 6 mg/kg for maintenance dose via IV infusion every 3 weeks.
  Paclitaxel: 175 mg/m2 BSA via IV infusion on the day following the first dose of study drug (CT-P6). Paclitaxel cycles were repeated every 3 weeks.
- Herceptin: Herceptin: 8 mg/kg for loading or 6 mg/kg for maintenance dose via IV infusion every 3 weeks.
  Paclitaxel: 175 mg/m2 BSA via IV infusion on the day following the first dose of study drug (Herceptin). Paclitaxel cycles were repeated every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | CT-P6 | Herceptin | Total
Number analyzed (Participants) | 244 | 231 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (9.70) | 51.9 (10.75) | 52.9 (10.26)
Age, Customized [Count of Participants; unit: Participants]
  >=65 years | 34 | 22 | 56
  <65 years | 210 | 209 | 419
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 231 | 475
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 158 | 141 | 299
  Asian | 86 | 90 | 176
Region of Enrollment [Count of Participants; unit: Participants]
  Belarus | 8 | 8 | 16
  Bulgaria | 13 | 7 | 20
  Georgia | 10 | 11 | 21
  Hong Kong | 0 | 2 | 2
  India | 31 | 35 | 66
  South Korea | 31 | 32 | 63
  Latvia | 7 | 6 | 13
  Malaysia | 2 | 3 | 5
  Philippines | 17 | 15 | 32
  Poland | 4 | 4 | 8
  Romania | 6 | 7 | 13
  Russia | 47 | 39 | 86
  Serbia | 4 | 5 | 9
  Singapore | 1 | 0 | 1
  Thailand | 4 | 3 | 7
  Turkey | 4 | 2 | 6
  Ukraine | 55 | 52 | 107
Childbearing Potential [Count of Participants; unit: Participants]
  Yes | 53 | 74 | 127
  No | 191 | 157 | 348
Height at Screening [Mean (Standard Deviation); unit: cm] | 159.5 (6.98) | 158.9 (7.21) | 159.2 (7.09)
Weight at Screening [Mean (Standard Deviation); unit: kg] | 67.5 (14.85) | 69.3 (16.06) | 68.4 (15.46)
BSA at Screening [Mean (Standard Deviation); unit: m2] | 1.72 (0.203) | 1.74 (0.220) | 1.73 (0.212)
Prior Chemotherapy [Count of Participants; unit: Participants]
  Yes | 107 | 100 | 207
  No | 137 | 131 | 268
ECOG performance status [Count of Participants; unit: Participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    Grade 0 | 128 | 116 | 244
    Grade 1 | 115 | 115 | 230
    Grade 2 | 1 | 0 | 1
Karnofsky performance status [Count of Participants; unit: Participants] — Category 1 (80-100 points): Able to carry on normal activity and to work; no special care needed.
  Category 2 (50-70 points): Unable to work; able to live at home and care for most personal needs; varying amount of assistance needed.
  Participants
    Category 1 | 236 | 217 | 453
    Category 2 | 4 | 7 | 11
    Not reported | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Best Overall Response (BOR) was derived from the overall response across all time points until after Cycle 8 using Independent Tumor Review Committee (ITRC) data in the FAS. Objective Response Rate (ORR) was defined as the number of patients with a BOR of complete response (CR) or partial response (PR) divided by the number of patients in the corresponding population, as assessed by Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1.
Time Frame: 6 months (up to 24 weeks)
Population: Full Analysis Set - consisted of all randomized patients who received any study drug and had at least one post-baseline assessment, with the exception of the patients who violated against Herceptin indication.
  All outcome measures of the Phase 3 study (CT-P6 3.1) were analyzed in conjunction with those of the Phase 1/2b study (CT-P6 1.1).
Measure: Count of Participants; unit: Participants
Groups:
- CT-P6: The ORR results for CT-P6 treatment group based on BOR during the Main Study Treatment Period (up to Cycle 8; 6 months) from the ITRC are presented below.
- Herceptin: The ORR results for Herceptin treatment group based on BOR during the Main Study Treatment Period from the ITRC are presented below.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 244 | 231
Participants | 138 | 143
Statistical Analysis 1: Comparison: CT-P6 vs Herceptin; Test type: Equivalence — The therapeutic equivalence between CT-P6 and Herceptin is concluded if the 95% confidence interval (CI) for the risk difference (CT-P6 - Herceptin) estimate in ORR ITRC review during the Main Study Treatment Period is entirely within the predefined equivalence margin of -0.15 to 0.15; Risk Difference (RD) = -0.0535, 95% CI 2-sided [-0.143 to 0.036]

2. Secondary Outcome: Time to Progression
Description: Time from randomization to determined progressive disease, as assessed by RECIST version 1.1.
Time Frame: Through study completion, approximately 40 months
Population: Full Analysis Set (FAS) - consisted of all randomized patients who received any study drug and had at least one post-baseline assessment, with the exception of the patients who violated against Herceptin indication.
  All outcome measures of the Phase 3 study (CT-P6 3.1) were analyzed in conjunction with those of the Phase 1/2b study (CT-P6 1.1).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CT-P6: The TTP results for CT-P6 treatment group in the FAS from the ITRC (up to 1 year) and from the Investigator are presented below.
- Herceptin: The TTP results for Herceptin treatment group in the FAS from the ITRC (up to 1 year) and from the Investigator are presented below.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 244 | 231
months
  ITRC | 11.07 [9.69 to 12.42] | 12.52 [11.10 to NA] — Not estimable due to insufficient number of event.
  Investigator | 10.99 [9.70 to 11.71] | 11.25 [9.74 to 12.47]

3. Secondary Outcome: Time to Response
Description: Time from randomization to observed tumor response (Complete Response or Partial Response), as assessed by RECIST 1.1
Time Frame: Through study completion, approximately 40 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CT-P6: The TTR results for CT-P6 treatment group in the FAS from the ITRC (up to 1 year) and from the Investigator are presented below.
- Herceptin: The TTR results for Herceptin treatment group in the FAS from the ITRC (up to 1 year) and from the Investigator are presented below.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 244 | 231
months
  ITRC | 1.38 [1.38 to 1.41] | 1.38 [1.38 to 1.41]
  Investigator | 1.41 [1.41 to 1.45] | 1.41 [1.38 to 1.45]

4. Secondary Outcome: Progression Free Survival
Description: Time from randomization to radiological progression or death from any cause, as assessed by RECIST 1.1
Time Frame: Through study completion, approximately 40 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CT-P6: The PFS results for CT-P6 treatment group in the FAS from the Investigator are presented below.
- Herceptin: The PFS results for Herceptin treatment group in the FAS from the Investigator are presented below.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 244 | 231
months | 10.99 [9.67 to 11.58] | 11.15 [9.74 to 12.43]

5. Secondary Outcome: Overall Survival
Description: The number of days between the date of randomization and the date of death from any cause.
Time Frame: Through study completion, approximately 40 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CT-P6: The OS results for CT-P6 treatment group in the FAS from the Investigator are presented below.
- Herceptin: The OS results for Herceptin treatment group in the FAS from the Investigator are presented below.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 244 | 231
months | 28.82 [25.10 to 32.96] | 26.84 [22.43 to 32.50]

6. Secondary Outcome: Safety Endpoints; Cardiotoxicity
Description: Mean change from baseline to endpoint assessment in left ventricular ejection fraction (LVEF) (%)
Time Frame: Through study completion, approximately 40 months
Population: Safety Analysis Set (SAF) - consisted of all patients in the FAS, analyzed as treated. All patients who received at least one dose of CT-P6 were analyzed under the CT-P6 treatment group. All other patients were analyzed under the Herceptin treatment group.
  All outcome measures of the Phase 3 study (CT-P6 3.1) were analyzed in conjunction with those of the Phase 1/2b study (CT-P6 1.1).
Measure: Mean (Standard Deviation); unit: %; percent change in LVEF
Groups:
- CT-P6: The mean change from baseline to worst value from the ITRC for CT-P6 treatment group is presented below.
- Herceptin: The mean change from baseline to worst value from the ITRC for Herceptin treatment group is presented below.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 185 | 173
%; percent change in LVEF | -4.56 (6.56) | -4.98 (6.54)

7. Secondary Outcome: Safety Endpoints; Immunogenicity
Description: Assessed by the proportion of patients with development of antibodies to study drug (positive anti-drug antibody [ADA] results after the first study drug infusion)
Time Frame: During treatment, median of 13 cycles (every cycle is 3 weeks)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- CT-P6: The immunogenicity results for CT-P6 treatment group are presented below.
- Herceptin: The immunogenicity results for Herceptin treatment group are presented below.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 244 | 231
Participants
  ADA positive patients with at least 1 result at any time during the study | 4 | 2
  ADA positive patients with a result at baseline visit: number analyzed (Participants) | 241 | 226
  ADA positive patients with a result at baseline visit | 1 | 2
  ADA positive patients with at least 1 result after the first infusion: number analyzed (Participants) | 235 | 218
  ADA positive patients with at least 1 result after the first infusion | 3 | 0

8. Secondary Outcome: Pharmacokinetic Endpoints; Ctroughss
Description: Trough concentration at steady state
Time Frame: predose and at 1.5 hours (end of infusion) of each cycle
Population: PK Analysis Set (PKAS) - consisted of all FAS patients who had achieved steady state by the 8th cycle, which required 3 consecutive similar trough concentrations.
  All outcome measures of the Phase 3 study (CT-P6 3.1) were analyzed in conjunction with those of the Phase 1/2b study (CT-P6 1.1).
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- CT-P6: The CtroughSS results for CT-P6 treatment group are presented below.
- Herceptin: The CtroughSS results for Herceptin treatment group are presented below.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 150 | 160
ug/mL | 23.6 (24.5) | 24.2 (27.8)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) reporting was extended from date of informed consent until completion of the final visit (up to approximately 57 months).
Description: At each level of summarization, patients were counted once if they reported one or more events.
Arm/Group | CT-P6 | Herceptin
All-Cause Mortality (participants affected / at risk) | 8/244 | 8/231
Serious Adverse Events (participants affected / at risk) | 34/244 | 39/231
Other Adverse Events (participants affected / at risk) | 227/244 | 214/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P6 (N=244) | Herceptin (N=231)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2)
Disease progression (General disorders) | 4 (4) | 6 (6)
Inflammation (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (3)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (3) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Endoscopic retrograde cholangiopancreatography (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulval ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Biliary drainage (Surgical and medical procedures) | 0 (0) | 1 (4)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Extended radical mastectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Mastectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P6 (N=244) | Herceptin (N=231)
Anaemia (Blood and lymphatic system disorders) | 31 (58) | 38 (67)
Leukopenia (Blood and lymphatic system disorders) | 28 (40) | 50 (85)
Neutropenia (Blood and lymphatic system disorders) | 68 (126) | 76 (156)
Abdominal pain (Gastrointestinal disorders) | 14 (20) | 13 (14)
Constipation (Gastrointestinal disorders) | 10 (14) | 18 (22)
Diarrhoea (Gastrointestinal disorders) | 34 (52) | 44 (74)
Nausea (Gastrointestinal disorders) | 41 (152) | 40 (75)
Stomatitis (Gastrointestinal disorders) | 14 (25) | 17 (20)
Vomiting (Gastrointestinal disorders) | 23 (34) | 27 (37)
Asthenia (General disorders) | 50 (132) | 34 (52)
Chills (General disorders) | 10 (15) | 19 (20)
Fatigue (General disorders) | 30 (78) | 34 (64)
Oedema peripheral (General disorders) | 10 (13) | 13 (18)
Pain (General disorders) | 11 (17) | 16 (31)
Pyrexia (General disorders) | 23 (40) | 28 (44)
Upper respiratory tract infection (Infections and infestations) | 8 (12) | 14 (19)
Alanine aminotransferase increased (Investigations) | 23 (51) | 24 (54)
Aspartate aminotransferase increased (Investigations) | 17 (28) | 15 (28)
Blood alkaline phosphatase increased (Investigations) | 13 (18) | 11 (19)
Gamma-glutamyltransferase increased (Investigations) | 18 (39) | 12 (27)
Decreased appetite (Metabolism and nutrition disorders) | 19 (37) | 16 (30)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 (23) | 15 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (82) | 33 (125)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (20) | 20 (30)
Bone pain (Musculoskeletal and connective tissue disorders) | 24 (63) | 17 (30)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 13 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 47 (173) | 53 (167)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (36) | 31 (49)
Dizziness (Nervous system disorders) | 17 (24) | 24 (35)
Headache (Nervous system disorders) | 21 (26) | 35 (48)
Neuropathy peripheral (Nervous system disorders) | 65 (147) | 58 (135)
Paraesthesia (Nervous system disorders) | 15 (16) | 9 (18)
Peripheral sensory neuropathy (Nervous system disorders) | 50 (125) | 54 (85)
Insomnia (Psychiatric disorders) | 11 (18) | 16 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (34) | 22 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 10 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 122 (153) | 127 (151)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (14) | 18 (24)
Rash (Skin and subcutaneous tissue disorders) | 19 (27) | 15 (39)
Hypertension (Vascular disorders) | 10 (12) | 14 (19)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (31) | 15 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes